CLINICAL TRIAL: NCT06429995
Title: Standard Follow-up Program (SFP) for Breast Cancer Patients
Acronym: SFPMAMMA
Status: Enrolling by invitation | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: SFP MAMMA
Record Dates: First submitted 2023-09-22; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: Acute toxicity; Late toxicity; Prediction models
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy; Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiotherapy
  Other Names: chemoradiation

SUMMARY:
Motive:

In order to improve the treatment technique, a comprehensive follow-up program is needed to obtain all relevant patient, treatment and toxicity data from breast cancer patients.

Goal:to set-up and maintain a database containing treatment results in terms of tumor control, side effects, complications and patient-reported quality of life.

A standard database of patiënts receiving photon treatment will be created. These data are then linked to dose-volume data of radiotherapy, with the aim to build prediction models for both tumor control and toxicity after radio (chemo) therapy that can later be used for selecting patients for proton treatment.

To set-up and maintain a database containing treatment results in terms of tumor control, side effects, complications and patient-reported quality of life.

A standard database of patients receiving photon treatment will be created. These data are then linked to dose-volume data of radiotherapy, with the aim to build prediction models for both tumor control and toxicity after radio (chemo) therapy that can later be used for selecting patients for proton treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer Patients receiving a radiotherapy dose

Exclusion Criteria:

* Failure to comply with any of the inclusion criteria

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with breast cancer receiving radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Score of Acute toxicity | Before start of radiation therapy and during radiation therapy and at 2 weeks after last day of radiation therapy.
  Acute Toxicity is measured with Common Terminology Criteria for Adverse Events (CTCAE).
Score of Late toxicity | At one and two years after last day of radiation therapy.
  Late Toxicity is measured with Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Overall survival | At 2 weeks after last day of radiation therapy and thereafter yearly, anticipated average 5-10 years.
  Overall survival
Loco-regional tumor control | At 2 weeks after last day of radiation therapy and thereafter yearly, anticipated average 5-10 years.
  Loco-regional tumor control

OTHER OUTCOMES:
Hemoglobin (Hb) | Before start of radiation therapy
  Hb level (mmol/l) measured in blood
Hematocrit (Ht) | Before start of radiation therapy
  Ht levels (L/L) measured in blood
Leukocytes | Before start of radiation therapy
  Leukocytes + differential count (10E9/l) measured in blood
Creatinine | Before start of radiation therapy
  Creatinine levels (mmol/l) measured in blood
Estimated Glomerular filtration rate (eGFR) | Before start of radiation therapy
  eGFR calculated from creatinine levels (ml/min)
Urea | Before start of radiation therapy
  Urea levels (mmol/l) measured in blood
Hemoglobin A1c (HbA1c) | Before start of radiation therapy
  HbA1c levels (mmol/mol) measured in blood
Cholesterol | Before start of radiation therapy
  Cholesterol levels (mmol/L) measured in blood
High-densitiy-lipoprotein cholesterol (HDL cholesterol) | Before start of radiation therapy
  HDL cholesterol levels (mmol/L) measured in blood
Low-density-lipoprotein cholesterol (LDL cholesterol) | Before start of radiation therapy
  LDL cholesterol levels (mmol/L) measured in blood
Triglycerides | Before start of radiation therapy
  Triglycerides levels (mmol/L) measured in blood
High sensitive C-reactive protein (hsCRP) | Before start of radiation therapy
  HsCRP levels (mg/L) measured in blood
Thyroid stimulating hormone (TSH) | Before start of radiation therapy, 1 and 2 years after radiation therapy
  TSH levels (mU/L) measured in blood
Free Thyroxine-4 (FT4) | Before start of radiation therapy, 1 and 2 years after radiation therapy
  FT4 levels (pmol/L) measured in blood
Patient-rated Demographics measured with the baseline questionnaire on Demographics | Before start of radiation therapy
  Patient-rated demographics measured with the baseline questionnaire on Demographics (unvalidated questionnaire)
Patient-rated symptoms measured with the EORTC QLQ-BR23 | Before start of radiation therapy, at 2 weeks after last day of radiation therapy, and at 3,6,12 months after last day of radiation therapy and thereafter yearly, anticipated average 20 years
  Patient-rated symptoms are measured with the Quality of Life Questionnaire-BR23 (EORTC QLQ-BR23)
Patient-rated symptoms measured with the BCSCQ | Before start of radiation therapy, at 2 weeks after last day of radiation therapy, and at 3,6,12 months after last day of radiation therapy and thereafter yearly, anticipated average 20 years.
  Patient-rated symptoms are measured with the Breast Cancer Questionnaire (BCSCQ: Based on the BCTOS (1) and the questionnaire on Patients' satisfaction with the cosmetic outcome by Sneeuw at al.(2))
Patient-rated symptoms measured with the questionnaire on Cardiovascular Diseases and Risk Factors and Lung Diseases (baseline) | Before start of radiation therapy
  Patient-rated symptoms are measured with the baseline questionnaire on Cardiovascular Diseases and Risk Factors and Lung Diseases before start of radiation therapy (unvalidated questionnaire)
Patient-rated symptoms with the questionnaire on Cardiovascular Diseases and Risk Factors and Lung Diseases (follow up) | 6 and 12 months after last day of radiation therapy and thereafter yearly, anticipated average 20 years
  Patient-rated symptoms are measured with the follow up questionnaire on Cardiovascular Diseases and Risk Factors and Lung Diseases (semi)annually after last day of radiation therapy (unvalidated questionnaire)
Patient-rated symptoms measured with the questionnaire on Performance Status | Before start of radiation therapy, at 2 weeks after last day of radiation therapy, and at 3,6,12 months after last day of radiation therapy and thereafter yearly, anticipated average 20 years
  Patient-rated symptoms are measured with the questionnaire on Performance Status (unvalidated questionnaire)
: Patient-rated symptoms measured with the questionnaire on Locoregional Tumor Control/New Primary Tumor | 6 and 12 months after last day of radiation therapy and thereafter yearly, anticipated average 20 years
  Patient-rated symptoms are measured with the questionnaire on Locoregional Tumor Control/New Primary Tumor (unvalidated questionnaire)
Patient-rated Quality of Life measured with the EORTC QLQ-C30 | Before start of radiation therapy, at 2 weeks after last day of radiation therapy, and at 3,6,12 months after last day of radiation therapy and thereafter yearly, anticipated average 20 years
  Patient-rated quality of life is measured with the Quality-of-Life Questionnaire-C30 (EORTC QLQ-C30)
Patient-rated Quality of Life measured with the EuroQoL-5D_5L | Before start of radiation therapy, at 2 weeks after last day of radiation therapy, and at 3,6,12 months after last day of radiation therapy and thereafter yearly, anticipated average 20 years
  Patient-rated quality of life is measured with the EuroQol Health questionnaire 5-level version (EuroQoL-5D_5L)
Patient-rated Quality of Life measured with EORTC QLQ-BR23 | Before start of radiation therapy, at 2 weeks after last day of radiation therapy, and at 3,6,12 months after last day of radiation therapy and thereafter yearly, anticipated average 20 years
  Patient-rated quality of life is measured with the Quality of Life Questionnaire-BR23 (EORTC QLQ-BR23).

CONTACTS AND LOCATIONS:
Overall Officials: Anne Crijns, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Background] Stanton AL, Krishnan L, Collins CA. Form or function? Part 1. Subjective cosmetic and functional correlates of quality of life in women treated with breast-conserving surgical procedures and radiotherapy. Cancer. 2001 Jun 15;91(12):2273-81. PMID 11413515
- [Background] Sneeuw KC, Aaronson NK, Yarnold JR, Broderick M, Regan J, Ross G, Goddard A. Cosmetic and functional outcomes of breast conserving treatment for early stage breast cancer. 1. Comparison of patients' ratings, observers' ratings, and objective assessments. Radiother Oncol. 1992 Nov;25(3):153-9. doi: 10.1016/0167-8140(92)90261-r. PMID 1470691